CLINICAL TRIAL: NCT03807245
Title: A Phase I, Randomised, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Safety, Tolerability and Immunogenicity of Two Doses of Group B Streptococcus Vaccine (GBS-NN/NN2 With Alhydrogel®) in Healthy Female Subjects Aged 18 to 40
Brief Title: Group B Streptococcus Vaccine in Healthy Females
Acronym: MVX0002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Minervax ApS (Other)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-003871-27
Record Dates: First submitted 2019-01-09; First posted 2019-01-16 (Actual); Results first posted 2020-12-24 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2020-11

CONDITIONS: Group B Strep Infection
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GBS-NN/NN2 with Alhydrogel® 25 (Experimental): GBS-NN/NN2 with Alhydrogel® 25 mcg intramuscular 2 times with 4 weeks apart
  Interventions: Biological: GBS-NN/NN2 with Alhydrogel® 25
- Placebo GBS-NN/NN2 with Alhydrogel® 25 (Placebo Comparator): Intramuscular injection with Alhydrogel® 2 times with 4 weeks apart
  Interventions: Biological: Placebo GBS-NN/NN2 with Alhydrogel® 25
- GBS-NN/NN2 with Alhydrogel® 50 (Experimental): Intramuscular GBS-NN/NN2 with Alhydrogel® injection 50 mcg 2 times with 4 weeks apart
  Interventions: Biological: GBS-NN/NN2 with Alhydrogel® 50
- Placebo GBS-NN/NN2 with Alhydrogel® 50 (Placebo Comparator): Intramuscular injection with Alhydrogel® 2 times with 4 weeks apart
  Interventions: Biological: Placebo GBS-NN/NN2 with Alhydrogel® 50

INTERVENTIONS:
Biological: GBS-NN/NN2 with Alhydrogel® 25 — GBS-NN/NN2 with Alhydrogel® vaccine will administered to subjects intramuscular 2 times with 4 weeks apart
  Arms: GBS-NN/NN2 with Alhydrogel® 25
Biological: Placebo GBS-NN/NN2 with Alhydrogel® 25 — GBS-NN/NN2 with Alhydrogel® vaccine will administered to subjects intramuscular 2 times with 4 weeks apart
  Arms: Placebo GBS-NN/NN2 with Alhydrogel® 25
Biological: Placebo GBS-NN/NN2 with Alhydrogel® 50 — GBS-NN/NN2 with Alhydrogel® vaccine will administered to subjects intramuscular 2 times with 4 weeks apart
  Arms: Placebo GBS-NN/NN2 with Alhydrogel® 50
Biological: GBS-NN/NN2 with Alhydrogel® 50 — GBS-NN/NN2 with Alhydrogel® vaccine will administered to subjects intramuscular 2 times with 4 weeks apart
  Arms: GBS-NN/NN2 with Alhydrogel® 50

SUMMARY:
A Phase I, randomised, single centre, double-blind, placebo-controlled, parallel group study to evaluate the safety, tolerability and immunogenicity of two doses of Group B Streptococcus vaccine.

DETAILED DESCRIPTION:
There will be 4 arms in 2 cohorts of 30 subjects. Cohort 1 will receive two 0.5 mL injections, 4 weeks apart, each consisting of 25 μg of GBS-NN and 25 μg of GBS-NN2 (24 subjects) or placebo (6 subjects). Cohort 2 (30 subjects) will receive two 0.5 mL injections, 4 weeks apart, each consisting of 50 μg of GBS-NN and 50 μg of GBS-NN2 (24 subjects) or placebo (6 Subjects). All vaccines will be adsorbed to 500 μg Al3+ as Alhydrogel®.

Safety will be assessed after all subjects have completed Visit 4 (Day 8) for Cohort 1, at which point the decision will be made as to whether proceeding with administration of the doses in cohort 2 is appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects aged 18 - 40 years.
2. Body mass index (BMI) ≥18 and ≤30 kg/m2.
3. Subjects weight ≥50kg and ≤100kg at screening.
4. Able to voluntarily provide written informed consent to participate in the study.
5. Subjects are pre-menopausal.
6. Females of childbearing potential must have a negative pregnancy test at screening (β HCG) and prior to each dose. To prevent pregnancy female subjects of childbearing potential must take adequate contraceptive precautions for the entire duration of study participation (up to Day 85). Adequate and highly effective contraceptive precautions include:

   * Established use of oral, injected or implanted hormonal methods of contraception.
   * Placement of an intrauterine device (IUD) or intrauterine system (IUS).
   * Barrier methods of contraception: Condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
   * Male sterilisation (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). [For female subjects, the vasectomised male partner should be the sole partner for that subject].
   * True abstinence, when this is in line with the preferred and usual lifestyle of the subject.

   [Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception].

   • The chosen contraception method(s) must be followed from the first dose until at least Day 85 of the study.
7. Non-smokers for at least 3 months prior to first study vaccine administration.

Exclusion Criteria:

1. Subjects who have received GBS-NN vaccine previously.
2. Subjects with history or presence of significant cardiovascular disease, pulmonary, hepatic, gallbladder or biliary tract, renal, haematological, gastrointestinal, endocrine, immunologic, dermatological, neurological, psychiatric, autoimmune disease or current infection.
3. Pregnant or lactating females.
4. Laboratory values at screening which are deemed by the investigator to be clinically significantly abnormal.
5. Positive drug screen for drugs of abuse or a positive alcohol urine test prior to first dosing unless there is a documented medical explanation for the positive result other than drugs of abuse (e.g., the subject has been prescribed opioids for pain).
6. Positive for human immunodeficiency virus (HIV), hepatitis B or hepatitis C.
7. Participation in a clinical drug study during the 90 days preceding the initial dose in this study.
8. Any significant illness during the 4 weeks preceding check-in for this study (Day 1).
9. Subjects with a history of allergic reactions after previous vaccination.
10. Subjects who have received any vaccine within 30 days of screening, or who are planning to receive a vaccine up to Day 85 of the study.
11. Subjects receiving immunosuppressive therapy in the 6 months prior to screening, taking any short-term medications including over-the-counter (OTC) preparations, within 7 days of the first dose. Chronic medications such as antihypertensives, bronchodilators, oral contraceptives or statins that do not affect the immune system, will be permitted and allowed to continue during the study at the discretion of the Investigator. Paracetamol will be permitted for the treatment of headache or other symptoms. Use of OTC vitamins and dietary supplements is allowed
12. Subjects with tattoos at the proposed site of vaccine administration.
13. Donation of blood or blood products within 90 days prior to vaccine administration or intending to donate blood or blood products within 90 days of the last visit.
14. Subjects who, in the opinion of the Investigator, are unsuitable for participation in the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2020-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Kitson, Study Director — gkitson@propharmapartners.uk.com
Locations (1):
- Simbec Research Limited, Merthyr Tydfil, Wales, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy female participants aged 18 to 40 years were recruited in a Phase 1 unit from January 2019 and the study was completed by October 2019.
Groups:
- GBS-NN/NN2 With Alhydrogel® 25: GBS-NN/NN2 with Alhydrogel® containing 25 mcg of each GBS-NN and GBS-NN2 administered by intramuscular injection 2 times with 4 weeks apart
- GBS-NN/NN2 With Alhydrogel® 50: GBS-NN/NN2 with Alhydrogel® containing 50 mcg of each GBS-NN and GBS-NN2 administered by intramuscular injection 2 times with 4 weeks apart
- Placebo With Alhydrogel®: Placebo (buffer with Alhydrogel®) vaccine administered by intramuscular injection 2 times with 4 weeks apart
Period: Overall Study
Arm/Group | GBS-NN/NN2 With Alhydrogel® 25 | GBS-NN/NN2 With Alhydrogel® 50 | Placebo With Alhydrogel®
Started | 24 | 24 | 12
Completed | 23 | 24 | 12
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GBS-NN/NN2 With Alhydrogel® 25 | GBS-NN/NN2 With Alhydrogel® 50 | Placebo With Alhydrogel® | Total
Number analyzed (Participants) | 24 | 24 | 12 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.8 (5.36) | 30.8 (6.04) | 27.3 (5.53) | 29.7 (5.72)
Sex: Female, Male [Count of Participants; unit: Participants] — Healthy females
  Participants
    Female | 24 | 24 | 12 | 60
    Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 24 | 12 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 23 | 24 | 12 | 59
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 24 | 24 | 12 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Number of Participants with Treatment Emergent Adverse Events
Time Frame: 85 days
Measure: Count of Participants; unit: Participants
Groups:
- GBS-NN/NN2 With Alhydrogel® 50: GBS-NN/NN2 with Alhydrogel® containing 50mcg of each GBS-NN and GBS-NN2 administered by intramuscular injection 2 times with 4 weeks apart
- Placebo With Alhydrogel®: Placebo (buffer with Alhydrogel®) administered by intramuscular injection 2 times with 4 weeks apart
Arm/Group | GBS-NN/NN2 With Alhydrogel® 25 | GBS-NN/NN2 With Alhydrogel® 50 | Placebo With Alhydrogel®
Number analyzed (Participants) | 24 | 24 | 12
Participants | 17 | 15 | 8

2. Secondary Outcome: Immunoglobulin(Ig)G Antibody Concentration
Description: Adjusted geometric mean concentration (GMC)
Time Frame: Day 85
Measure: Geometric Mean (95% Confidence Interval); unit: Adjusted GMC mcg/mL
Arm/Group | GBS-NN/NN2 With Alhydrogel® 25 | GBS-NN/NN2 With Alhydrogel® 50 | Placebo With Alhydrogel®
Number analyzed (Participants) | 24 | 24 | 12
Adjusted GMC mcg/mL
  GBS-NN | 15.2 [11.1 to 20.8] | 17.1 [12.5 to 23.4] | 0.115 [0.0746 to 0.177]
  GBS-NN2 | 24.0 [18.8 to 30.8] | 29.9 [23.4 to 38.3] | 0.154 [0.109 to 0.216]

3. Secondary Outcome: Fold Change in Antibody Concentration
Description: Geometric mean fold change in antibody concentration from Day 1 to Day 85 for each group.
Time Frame: Day 1 to Day 85
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change from Day 1 to Day 85
Arm/Group | GBS-NN/NN2 With Alhydrogel® 25 | GBS-NN/NN2 With Alhydrogel® 50 | Placebo With Alhydrogel®
Number analyzed (Participants) | 24 | 24 | 12
Fold change from Day 1 to Day 85
  GBS-NN | 127.707 [79.310 to 205.637] | 131.526 [93.987 to 184.057] | 0.951 [0.791 to 1.144]
  GBS-NN2 | 169.594 [104.224 to 275.964] | 211.303 [140.290 to 318.260] | 0.946 [0.838 to 1.068]
Statistical Analysis 1: Comparison: GBS-NN/NN2 With Alhydrogel® 25 vs Placebo With Alhydrogel®; Adjusted geometric mean fold increase from Day 1 to Day 85: adjusted geometric mean ratio GBS-NN/NN2 25mcg/placebo; Test type: Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: GBS-NN/NN2 With Alhydrogel® 50 vs Placebo With Alhydrogel®; Adjusted geometric mean fold increase from Day 1 to Day 85: adjusted geometric mean ratio GBS-NN/NN2 50mcg/placebo; Test type: Other; p < 0.0001, ANOVA

4. Secondary Outcome: Seroconversion Rate
Description: 4-fold increase in Immunoglobulin(Ig)G antibody concentration
Time Frame: Day 85
Measure: Count of Participants; unit: Participants
Arm/Group | GBS-NN/NN2 With Alhydrogel® 25 | GBS-NN/NN2 With Alhydrogel® 50 | Placebo With Alhydrogel®
Number analyzed (Participants) | 23 | 23 | 12
Participants
  GBS-NN | 23 | 23 | 0
  GBS-NN2 | 23 | 23 | 0

5. Secondary Outcome: Number of Participants With an Immune Response to First and Second Doses
Description: Number of participants with Immunoglobulin(Ig)G antibody concentration above thresholds
Time Frame: Day 29 and Day 85
Measure: Count of Participants; unit: Participants
Arm/Group | GBS-NN/NN2 With Alhydrogel® 25 | GBS-NN/NN2 With Alhydrogel® 50 | Placebo With Alhydrogel®
Number analyzed (Participants) | 24 | 24 | 12
Participants
  GBS-NN Day 29 increase above 1mcg/mL | 19 | 23 | 0
  GBS-NN Day 29 increase above 2mcg/mL | 19 | 20 | 0
  GBS-NN Day 29 increase above 4mcg/mL | 17 | 17 | 0
  GBS-NN Day 29 increase above 8mcg/mL | 13 | 13 | 0
  GBS-NN Day 85 increase above 1mcg/mL | 23 | 23 | 0
  GBS-NN Day 85 increase above 2mcg/mL | 20 | 23 | 0
  GBS-NN Day 85 increase above 4mcg/mL | 20 | 21 | 0
  GBS-NN Day 85 increase above 8mcg/mL | 18 | 20 | 0
  GBS-NN2 Day 29 increase above 1mcg/mL | 20 | 22 | 0
  GBS-NN2 Day 29 increase above 2mcg/mL | 18 | 22 | 0
  GBS-NN2 Day 29 increase above 4mcg/mL | 17 | 18 | 0
  GBS-NN2 Day 29 increase above 8mcg/mL | 16 | 18 | 0
  GBS-NN2 Day 85 increase above 1mcg/mL | 23 | 23 | 0
  GBS-NN2 Day 85 increase above 2mcg/mL | 22 | 22 | 0
  GBS-NN2 Day 85 increase above 4mcg/mL | 20 | 22 | 0
  GBS-NN2 Day 85 increase above 8mcg/mL | 18 | 22 | 0

ADVERSE EVENTS:
Time Frame: 85 days
Arm/Group | GBS-NN/NN2 With Alhydrogel® 25 | GBS-NN/NN2 With Alhydrogel® 50 | Placebo With Alhydrogel®
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/12
Other Adverse Events (participants affected / at risk) | 17/24 | 15/24 | 8/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GBS-NN/NN2 With Alhydrogel® 25 (N=24) | GBS-NN/NN2 With Alhydrogel® 50 (N=24) | Placebo With Alhydrogel® (N=12)
Palpitations (Cardiac disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 2 | 1 | 0
Allergy to animal (Immune system disorders) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 2 | 2
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 2 | 0 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 9 | 5 | 5
Lethargy (Nervous system disorders) | 1 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 1 | 0
Hypomenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/45/NCT03807245/Prot_SAP_000.pdf